CLINICAL TRIAL: NCT04137029
Title: Effect of Methacholine, Long-acting M-cholinolytic and beta2-agonist on the Binding Activity of Beta-receptors in Healthy Volunteers
Brief Title: Methacholine, Long-acting M-cholinolytic and beta2-agonist on the Activity of Beta-receptors in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, Pulmonology Scientific Research Institute (Other Government)
Collaborators: Moscow State University of Medicine and Dentistry (Other); National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government); Branch of Shemyakin-Ovchinnikov Institute of Bioorganic chemistry of RAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PSRI04-19
Record Dates: First submitted 2019-10-11; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Health, Subjective; Hyperreactivity, Bronchial
Keywords: beta-receptors; metacholine; formoterol; tiotropium
MeSH Terms: conditions — Bronchial Hyperreactivity | interventions — Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: There are two groups: the first group is smokers, the second group is non - smokers. The participants of both groups will receive metacholine on the first visit, formoterol 12 micrograms on the second visit, then tiotropium bromide 18 mkg on the third visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoking (Experimental): Healthy smoking volunteers
  Interventions: Drug: Formoterol; Drug: Tiotropium Bromide; Diagnostic Test: metacholine test
- non-smoking (Experimental): Healthy non-smoking volunteers
  Interventions: Drug: Formoterol; Drug: Tiotropium Bromide; Diagnostic Test: metacholine test

INTERVENTIONS:
Drug: Formoterol — The participants will receive inhalation of formoterol 12 micrograms
Drug: Tiotropium Bromide — The participants will receive inhalation of tiotropium bromide 18 mkg once
Diagnostic Test: metacholine test — The participants will receive inhalation of metacholine once

SUMMARY:
Interventional open-labeled study in parallel groups is aimed to evaluate changes of beta receptors in healthy volunteers under the influence of inhaled metacholine, long-acting anticholinergics and beta-agonists using modified radioligand method.

DETAILED DESCRIPTION:
Long-acting beta2-agonists and anticholinergics are main drugs in therapy of chronic obstructive pulmonary disease . Beta-agonists exert their bronchodilatory effects via β2 adrenoceptors located on airway smooth muscle cells. Anticholinergics block mainly M3-cholinoreceptors located in the airways, thus inhibiting bronchoconstriction. Metacholine blocks M2-cholinoreceptors thus inducing bronchoconstriction. It is known, that muscarine and beta-receptors interact with each other, but the detailed mechanism is unknown. For evaluating the binding activity of beta-receptors after inhalation of these drugs the modified radioligand method was used.

ELIGIBILITY:
Inclusion Criteria:

1 Provision of signed and dated informed consent form 2. Healthy male or female, aged 18-60 years

Exclusion Criteria:

* Participants unable to perform spirometry
* Exacerbation respiratory infection within the previous four weeks
* Hypersensitivity or allergy to formoterol, metacholine or tiotropium bromide
* Females who are currently pregnant and lactating
* major surgery in the last 6 months
* Refusal to participate
* Currently participating in another clinical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline beta-receptor binding activity at 60 min after the inhalation of formoterol or tiotropium. | Baseline (pre-dose), 60 minutes
  Beta-receptor binding activity will be measured with modified radioligand method before and after 60 min after the inhalation of formoterol or tiotropium
Change from baseline beta-receptor binding activity at 40 min after the challenge test with metacholine. | Baseline (pre-dose), 40 minutes
  Beta-receptor binding activity will be measured with modified radioligand method before and after 40 min after the challenge test with metacholine.

SECONDARY OUTCOMES:
Comparison of beta-receptor binding activity measured with modified radioligand after formoterol and tiotropium. | Baseline (pre-dose), 60 minutes
  Difference of change of beta-receptor binding activity measured with modified radioligand method before and after 60 min after the inhalation of formoterol and tiotropium.
Comparison of beta-receptor binding activity measured with modified radioligand method after formoterol or tiotropium in smokers and non-smokers. | Baseline (pre-dose), 60 minutes
  Difference of change of beta-receptor binding activity measured with modified radioligand method before and after 60 min after the inhalation of formoterol or tiotropium in smokers and non-smokers.
Comparison of beta-receptor binding activity measured with modified radioligand after metacholine | Baseline (pre-dose), 40 minutes
  Difference of change of beta-receptor binding activity measured with modified radioligand method before and after inhalation of metacholine
Comparison of beta-receptor binding activity measured with modified radioligand method after inhalation of metacholine in smokers and non-smokers. | Baseline (pre-dose), 40 minutes
  Difference of change of beta-receptor binding activity measured with modified radioligand method before and after inhalation of metacholine

CONTACTS AND LOCATIONS:
Overall Officials: Kirill A Zykov, Prof, Principal Investigator — Federal State Budgetary Institution, Pulmonology Scientific Research Institute
Locations (1):
- Kirill Zykov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agapova OY, Skoblov YS, Zykov KA, Rvacheva AV, Beilina VB, Masenko VP, Chazova IE. [Radioligand Method of Assessment of beta-Adrenoceptor's Activity on Human T-Lymphocytes]. Bioorg Khim. 2015 Sep-Oct;41(5):592-8. doi: 10.1134/s1068162015050027. Russian. PMID 26762097
- [Result] Agapova OY, Skoblov YS, Tkachev GA, Mironova NA, Golitsyn SP, Masenko VP, Chazova IE, Zykov KA. [Changes in the receptor activity of beta2-adrenoreceptors of human T-lymphocytes under the effect of beta2-agonists]. Mol Biol (Mosk). 2016 Nov-Dec;50(6):999-1006. doi: 10.7868/S0026898416050025. Russian. PMID 28064316
- [Result] Smolyakova E.V., Skoblov Y.S., Skoblova N.A., Agapova O.Y., Ambat'ello L.G., Klimova A.A., Kuznetsova T.V., Masenko V.P., Nistor S.Yu., Rvacheva A.V., Chazova I.E., Zykov K.A. Specificity and Selectivity of the Modified Radioligand Method for Assessment of β1-Adrenoreceptor's Binding Activity on Human T-Lymphocytes. Russian Journal of Bioorganic Chemistry 45(3): 295-301, 2019